CLINICAL TRIAL: NCT02147769
Title: Cerebral Oxygenation and Autoregulation in Preterm Infants: Association With Morbidity and Mortality
Brief Title: Cerebral Oxygenation and Autoregulation in Preterm Infants
Acronym: Early NIRS
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Valerie Chock, M.D., M.S. Epi, Principle Investigator, Stanford University
Other Study IDs: 23894
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Intraventricular Hemorrhage of Prematurity; Complications of Prematurity
Keywords: cerebral autoregulation; preterm; near-infrared spectroscopy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants monitored with NIRS: All infants enrolled in the study will be monitored with cerebral near-infrared spectroscopy (NIRS monitoring) to measure cerebral oxygenation levels in the first 96 hours of life. Mean arterial blood pressure will simultaneously be monitored.
  Interventions: Device: NIRS monitoring

INTERVENTIONS:
Device: NIRS monitoring — All enrolled infants will undergo NIRS monitoring of cerebral oxygenation in addition to monitoring of continuous arterial blood pressure.

SUMMARY:
Premature infants are at high risk for variations in blood pressure and oxygenation during the first few days of life. The immaturity of the premature brain may further predispose these infants to death or the development of neurologic problems. The relationship between unstable blood pressure and oxygen levels and brain injury has not been well elucidated.

This study investigates the utility of near-infrared spectroscopy (NIRS), a non-invasive oxygen-measuring device, to identify preterm infants at highest risk for brain injury or death.

ELIGIBILITY:
Inclusion Criteria:

* inborn
* birth weight <= 1250 grams
* indwelling arterial catheter in place
* age <24 hours old

Exclusion Criteria:

* lethal chromosomal abnormality
* major congenital anomaly
* skin integrity insufficient to allow placement of NIRS sensors
* decision to not provide full intensive care

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All inborn preterm infants with birth weight <=1250 grams and with an indwelling arterial catheter already in place are eligible for study enrollment if they are <24 hours old at the time of enrollment. These preterm infants are at risk for impaired cerebral autoregulation and may undergo non-invasive monitoring of cerebral oxygenation using near-infrared spectroscopy (NIRS).
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Chock, MD, Principal Investigator — Stanford University; Krisa Van Meurs, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - St. John's Children's Hospital, Springfield, Illinois
  - Nationwide Children's Hospital, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Verhagen EA, Hummel LA, Bos AF, Kooi EM. Near-infrared spectroscopy to detect absence of cerebrovascular autoregulation in preterm infants. Clin Neurophysiol. 2014 Jan;125(1):47-52. doi: 10.1016/j.clinph.2013.07.001. Epub 2013 Aug 22. PMID 23973384
- [Background] Alderliesten T, Lemmers PM, Smarius JJ, van de Vosse RE, Baerts W, van Bel F. Cerebral oxygenation, extraction, and autoregulation in very preterm infants who develop peri-intraventricular hemorrhage. J Pediatr. 2013 Apr;162(4):698-704.e2. doi: 10.1016/j.jpeds.2012.09.038. Epub 2012 Nov 6. PMID 23140883
- [Background] Soul JS, Hammer PE, Tsuji M, Saul JP, Bassan H, Limperopoulos C, Disalvo DN, Moore M, Akins P, Ringer S, Volpe JJ, Trachtenberg F, du Plessis AJ. Fluctuating pressure-passivity is common in the cerebral circulation of sick premature infants. Pediatr Res. 2007 Apr;61(4):467-73. doi: 10.1203/pdr.0b013e31803237f6. PMID 17515873
- [Background] Wong FY, Silas R, Hew S, Samarasinghe T, Walker AM. Cerebral oxygenation is highly sensitive to blood pressure variability in sick preterm infants. PLoS One. 2012;7(8):e43165. doi: 10.1371/journal.pone.0043165. Epub 2012 Aug 14. PMID 22905222
- [Background] Caicedo A, De Smet D, Naulaers G, Ameye L, Vanderhaegen J, Lemmers P, Van Bel F, Van Huffel S. Cerebral tissue oxygenation and regional oxygen saturation can be used to study cerebral autoregulation in prematurely born infants. Pediatr Res. 2011 Jun;69(6):548-53. doi: 10.1203/PDR.0b013e3182176d85. PMID 21364491
- [Background] Wong FY, Leung TS, Austin T, Wilkinson M, Meek JH, Wyatt JS, Walker AM. Impaired autoregulation in preterm infants identified by using spatially resolved spectroscopy. Pediatrics. 2008 Mar;121(3):e604-11. doi: 10.1542/peds.2007-1487. Epub 2008 Feb 4. PMID 18250118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preterm Infants Monitored With NIRS
Started | 111
Completed | 111
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Preterm Infants Monitored With NIRS
Number analyzed (Participants) | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 111
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks gestational age] | 26 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 18
  White | 56
  More than one race | 5
  Unknown or Not Reported | 0
Death or Neuroradiographic abnormality at baseline [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Mortality Before Hospital Discharge
Description: Participants will be followed for the outcome of death prior to hospital discharge.
Time Frame: Outcome measure will be assessed at the time of subject's initial discharge from the hospital (on average by 40 weeks postmenstrual age), but at a maximum of 1 year of life.
Measure: Count of Participants; unit: Participants
Arm/Group | Preterm Infants Monitored With NIRS
Number analyzed (Participants) | 111
Participants | 11

2. Primary Outcome: Severe Central Nervous System (CNS) Morbidity
Description: Routine cranial ultrasound obtained within the first ten days of life will be utilized to detect grade 3 or 4 intraventricular hemorrhage, periventricular leukomalacia, significant ventriculomegaly, or white matter abnormalities.
Time Frame: Outcome measure will be assessed on day 10 of life. Participants will be followed for neuroradiographic evidence of CNS morbidity in the first ten days of life
Measure: Count of Participants; unit: Participants
Arm/Group | Preterm Infants Monitored With NIRS
Number analyzed (Participants) | 111
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse events were collected until hospital discharge or 6 months (whichever occurred first).
Arm/Group | Preterm Infants Monitored With NIRS
All-Cause Mortality (participants affected / at risk) | 11/111
Serious Adverse Events (participants affected / at risk) | 14/111
Other Adverse Events (participants affected / at risk) | 0/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preterm Infants Monitored With NIRS (N=111)
CNS abnormality (Nervous system disorders) | 14 (14) — Neuroradiographic abnormality on cranial ultrasound

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02147769/Prot_SAP_000.pdf